CLINICAL TRIAL: NCT05936112
Title: Quantification of Fecal Calprotectin Concentration Difference Between Infants Aged Under 4 Months Old Suffering From Functional Gastrointestinal Disorders (FGID) and Infants Aged Under 4 Months Old Free From Disorders : a Transversal Case-control Monocentric Study in Besançon
Brief Title: Quantification of Fecal Calprotectin Concentration Difference Between Infants Aged Under 4 Months Old Suffering From Functional Gastrointestinal Disorders (FGID) and Infants Aged Under 4 Months Old Free From Disorders : a Transversal Case-control Monocentric Study
Acronym: Cal-IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/793
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Functional Gastrointestinal Disorders; Infant, Newborn, Diseases
MeSH Terms: conditions — Gastrointestinal Diseases; Infant, Newborn, Diseases | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infants < 4 months old with FGID (Other): Infants < 4 months old presenting one or several Functional GastroIntestinal Disorder(s)
  Interventions: Other: Fecal calprotectin dosage; Other: Questionnaire and interview with parents
- Infants < 4 months old free from FGID (Other): Infants < 4 months old without any Functional GastroIntestinal Disorder
  Interventions: Other: Fecal calprotectin dosage; Other: Questionnaire and interview with parents

INTERVENTIONS:
Other: Fecal calprotectin dosage — Dosing calprotectin in infants' feces + questionnaire/interview with parents
Other: Questionnaire and interview with parents — Dosing calprotectin in infants' feces + questionnaire/interview with parents

SUMMARY:
There is a high prevalence of FGID among infants : 30 % for regurgitations, 20 % for colitis , 15 % for functional constipation.This represents a frequent motive for pediatrics consultation : 23 to 28 % of medical consultations in this population are consequent to gastrointestinal symptoms among infants aged under 4 months old. This can lead to numerous inappropriate or unrecommended medication prescriptions.

Currently, fecal calprotectin threshold are only validated by science societies for children aged 5 years old and more. This study aims to quantify the difference of fecal calprotectin between a population of infants for whom no FGID has been finally detected, and a population of infants for whom FGID have been detected during the gastro-pediatrics consultation, , in order to later determine wether it is possible to validate a threshold in a population of infants aged under 4 months old.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged under 4 months old benefiting from a special gastro-pediatrics consultation
* FGID arm : infant with one or several FGID detected
* Free from FGID arm : infant without any FGID detected

Exclusion Criteria:

* Born before 37 week of amenorrhea.
* Neurologic failure, heart failure, respiratory failure, hepatic failure, pancreatic failure, renal failure, cancer or hematological malignancy.
* History of enteral feeding by tube (nasogastric, nasojejunal, gastrostomy, gastrostomy-jejunostomy, jejunostomy) or parenteral feeding.
* History of digestive tract surgery
* Suspicion of Immunoglobulin E-mediated Cow's Milk Protein Allergy (CMPA): anaphylactic-type reaction observed within a few minutes to 2 hours after ingestion of cow's milk protein, such as pruritus, erythema, angioedema, intense abdominal pain, projectile vomiting, acute diarrhea, bronchospasm, faintness, loss of consciousness, arterial hypotension or even anaphylactic shock.

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Quantification of fecal calprotectin concentration difference | 1 month
  Quantification in µg/g feces of fecal calprotectin concentration difference between infants aged under 4 months old suffering from Functional Gastrointestinal disorders (FGID) and infants aged under 4 months old free from disorders

CONTACTS AND LOCATIONS:
Overall Officials: Eva OTT, MD, Principal Investigator — CHU de Besançon

IPD SHARING:
Plan to Share IPD: No